CLINICAL TRIAL: NCT01200563
Title: Comparative, Prospective, Randomized Study of MIST Therapy vs NPWT vs MIST Therapy in Conjunction With NPWT on the Rate of Healing and Its Economic Value in the Treatment of Full Thickness Wounds in a LTACH and SNF
Brief Title: Comparative Effectiveness Study of MIST Therapy Versus Negative Pressure Wound Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study site compliance
Sponsor: Celleration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-86000
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Wounds
Keywords: MIST Therapy; Negative Pressure Wound Therapy; Wound care in long-term acute care hospital; Wound care in skilled nursing facility setting
MeSH Terms: conditions — Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Subjects assigned to receive MIST Therapy will be treated 3 times per week. The duration of each MIST treatment will be dependent on the wound's area measured at baseline and at each weekly assessment.
  Interventions: Device: MIST Therapy
- Group 2 (Active Comparator): Subjects assigned to receive Negative Pressure Wound Therapy will be treated with the Vacuum Assisted Closure system. For administration of this study treatment, e.g., treatment cycle, target pressure and dressing changes, the manufacturer's recommended guidelines will be followed.
  Interventions: Device: Vacuum Assisted Closure
- Group 3 (Active Comparator): Subjects assigned to this group will receive MIST Therapy treatments and Negative Pressure Wound Therapy.
  Interventions: Device: MIST Therapy and Negative Pressure Wound Therapy

INTERVENTIONS:
Device: MIST Therapy — Low-frequency, non-contact ultrasound system delivering therapeutic ultrasound via a fine saline mist to the wound bed without direct contact of the device with the body.
  Other Names: MIST
  Arms: Group 1
Device: Vacuum Assisted Closure — Controlled negative pressure (vacuum) delivering negative (sub-atmospheric) pressure to the wound site applied by a tubing which decompresses a foam dressing, continuously or intermittently depending on wound type.
  Other Names: VAC Therapy
  Arms: Group 2
Device: MIST Therapy and Negative Pressure Wound Therapy — MIST Therapy will be provided 3 times per week, NPWT will be provided according to the manufacturer's recommended guidelines.
  Other Names: MIST; VAC Therapy
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the clinical and economic effectiveness of MIST Therapy vs NPWT vs MIST Therapy in conjunction with NPWT in the treatment of full thickness wounds presenting in the LTACH and SNF settings.

DETAILED DESCRIPTION:
A comparative, prospective, randomized study.

Study objectives: Comparison between study groups of the assigned study treatment's effect on the rate of wound healing, cost per episode of care, severity of wound pain, and the occurrence of adverse events.

Subject recruitment: Consecutive, prospective subjects admitted to the study site will be screened for study enrollment and potential randomization. Prospective data will be collected on study subjects until at least 10 subjects are randomized into each of three treatment groups: MIST Therapy; NPWT; or MIST Therapy and NPWT.

Protocol and procedures: All randomized subjects will continue to receive standard of care treatment appropriate for their wound for the duration of their study treatment regardless of their assigned treatment group. Subjects will continue to receive assigned study treatment as long as their wound continues to show improvement, as determined by the investigator. Study treatment will continue until wound closure, or for up to 6 weeks without wound closure. A baseline evaluation will include a medical history assessment, VAS pain score, wound history and evaluation including: wound dimension measurements, overall wound assessment, digital photography, and appropriate sharp debridement, if necessary. Weekly wound assessments will include a wound evaluation, digital photography and VAS pain score. Prospective data will also be collected on specific wound care supplies and interventions provided. These data will be tracked as interventions occur while the wound continues to be treated with the assigned study treatment. Economic data will include type, quantity, duration, associated frequency, and professional time requirements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of any race and at least 18 years old
* Subject presents with full thickness wound of any etiology
* Subject's wound is between 20cm2 and 250cm2
* Subject's wound has less that 20% necrotic tissue
* Subject is nutritionally stable and/or taking nutritional supplements and is being followed by a dietician
* Subject or subject's legally authorized representative understands the nature of the study procedure(s) and provides written informed consent prior to study enrollment
* Women of childbearing potential must not be pregnant or lactating, and must be using adequate and accepted contraceptive methods
* Subject has a reasonable expectation of completing the study
* Subject has had no prior MIST Therapy or Negative Pressure Wound Therapy to the enrolled wound

Exclusion Criteria:

* Subject's condition requires the use of topical antibiotics at the time of study enrollment
* Subject's wound would require ultrasound near an electronic implant or prosthesis, e.g., near or over the heart, or over the thoracic area if the patient is using a cardiac pacemaker
* Subject is known to be suffering from a disorder or other situation that the subject or investigator feels would interfere with compliance or other study requirements
* Subject is currently enrolled or has been enrolled in the last 30 days in another investigational device or drug trial
* Subject has a combination of medical condition(s) that in the opinion of the investigator would make the subject an inappropriate candidate for the study, i.e., diabetes, including renal, hepatic, hematologic, neurologic, or immune disease
* Subject's wound is not appropriate for Negative Pressure Wound Therapy or MIST Therapy
* Subject has osteomyelitis, systemic sepsis, or an infection not related to his/her index wound (e.g., UTI, pulmonary) that has been untreated or has not been appropriately managed
* Subject has a fistula(s) to the index wound bed
* Subject's index wound is a head or neck wound
* Subject's index wound presents with a malignancy in the wound bed
* Subject's anticoagulation therapy is unstable
* Subject is undergoing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Rate of wound healing. | 6 weeks
  Determined by the change in wound surface area/volume from the initial evaluation date to study end.

SECONDARY OUTCOMES:
Change wound exudation levels. | 6 weeks
  Determined by the change in amount of exudates recorded using a scale of none, mild, moderate, and heavy, from the initial evaluation date to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth O Anaeme, MD, Principal Investigator — Trillium Specialty Hospital
Locations (1):
- Trillium Specialty Hospital, Mesa, Arizona, United States